CLINICAL TRIAL: NCT04383561
Title: Leucin-rich alpha2 Glycoprotein (LRG): A Novel Acute Phase Protein Related With Stage 3 Periodontitis
Brief Title: Relationship Between LRG and Periodontal Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aydin Adnan Menderes University (Other)
Collaborators: Giresun University (Other); Bulent Ecevit University (Other)
Responsible Party: Principal Investigator, Zeynep Pinar KELES YUCEL, Assistant Prof., Giresun University
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: KAEK-92
Record Dates: First submitted 2020-05-04; First posted 2020-05-12 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2020-05

CONDITIONS: Periodontitis; Acute-Phase Response; Inflammation
Keywords: periodontitis; gingival crevicular fluid; serum
MeSH Terms: conditions — Periodontitis; Acute-Phase Reaction; Inflammation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- stage 3 periodontitis (Active Comparator): GCF and serum samples were collected before and after treatment from periodontitis patients.
  Interventions: Other: Non-surgical periodontal treatment; Other: Oral hygiene instructions
- Periodontally healthy controls (Placebo Comparator): GCF and serum samples were collected from periodontally healthy controls at baseline for once.
  Interventions: Other: Oral hygiene instructions

INTERVENTIONS:
Other: Non-surgical periodontal treatment — Scaling and root planing (SRP), in four clinical visits
  Arms: stage 3 periodontitis
Other: Oral hygiene instructions — Oral hygiene instructions includes brushing with the modified Bass technique, interdental cleaning with dental floss and interdental brushes.

SUMMARY:
This study aimed to investigate gingival crevicular fluid (GCF) and serum levels of LRG, interleukin (IL)-6 and tumor necrosis factor (TNF)-α in patients with periodontitis before and after non-surgical periodontal treatment.

DETAILED DESCRIPTION:
Twenty-five stage 3 periodontitis and twenty-five periodontally healthy individuals were enrolled in the study. Clinical periodontal measurements were recorded; periodontitis patients received non-surgical periodontal treatment, and GCF and serum samples were obtained at baseline and at 6 weeks after treatment. LRG, IL-6 and TNF-α were determined by ELISA.

ELIGIBILITY:
Inclusion Criteria:

1. 25-50 years of age
2. having at least 20 natural teeth, excluding third molars
3. having no systemic disease
4. non-smokers
5. criteria for healthy control group: BOP < 10% and PD ≤ 3 mm without clinical attachment loss or radiographic sign of alveolar bone destruction
6. criteria for stage 3 periodontitis group: interdental CAL ≥ 5 mm at least 2 non-adjacent teeth, PD ≥ 6 mm and radiographic bone loss extending to the mid-third of the root or beyond.

Exclusion Criteria:

1. having any systemic diseases,
2. smoking
3. current pregnancy or lactation
4. a history of periodontal treatment in the past 6 months
5. using antibiotic, anti-inflammatory drugs or any other drugs within the past 6 months.

Ages: 26 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2019-09-30 (Actual); Primary Completion 2020-01-15 (Actual); Study Completion 2020-02-15 (Actual)

PRIMARY OUTCOMES:
Changes in the levels of biochemical parameters | Baseline and 6 weeks after treatment
  The levels LRG, IL-6 and TNF-α were determined to define the diagnostic and prognostic potential as a biomarker in periodontitis.

CONTACTS AND LOCATIONS:
Locations (1):
- Giresun University, Giresun, Turkey (Türkiye)